CLINICAL TRIAL: NCT05683392
Title: Control-IQ 2.0 Feasibility Study #2: Use of Control-IQ Technology 2.0 in Adults, Children, and Preschoolers With Type 1 Diabetes
Brief Title: Use of Control-IQ Technology 2.0 in Adults, Children, and Preschoolers With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tandem Diabetes Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: TP-0011713
Record Dates: First submitted 2023-01-05; First posted 2023-01-13 (Actual); Results first posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes
Keywords: Control-IQ technology; type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Control-IQ 2.0 Lower Range First, then Standard Range (Experimental): After a two week run in period with Control-IQ 1.5, participants will use t:slim X2 pump with Control-IQ technology 2.0 with a lower range for two weeks, followed by use of t:slim X2 pump with Control-IQ technology 2.0 with a standard range for two weeks.
  Interventions: Device: t:slim X2 insulin pump with Control-IQ technology 2.0
- Control-IQ 2.0 Standard Range First, then Lower Range (Experimental): After a two week run in period with Control-IQ 1.5, participants will use t:slim X2 pump with Control-IQ technology 2.0 with a standard range for two weeks, followed by use of t:slim X2 pump with Control-IQ technology 2.0 with a lower range for two weeks.
  Interventions: Device: t:slim X2 insulin pump with Control-IQ technology 2.0

INTERVENTIONS:
Device: t:slim X2 insulin pump with Control-IQ technology 2.0 — t:slim X2 insulin pump with Control-IQ technology 2.0, and wearing the Dexcom G6 sensor.

SUMMARY:
The goal of this clinical trial is to assess safety of and explore glycemic outcomes with Control-IQ technology 2.0 in adults, children and preschoolers with type 1 diabetes.

DETAILED DESCRIPTION:
This feasibility study is a prospective, randomized, two-period crossover multi-center study of Control-IQ technology 2.0. After a two week run-in period, the automated insulin dosing (AID) system will be evaluated in multiple age groups over 4 weeks of use.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to ≤ 81 years
* Diagnosis of type 1 diabetes for at least 1 year, or at least 6 months for age 2-5 years at enrollment
* Prior Dexcom CGM user, with at least 11 of the prior 14 days of CGM use available for download at the screening visit to confirm eligibility
* Total Daily Insulin Dose (TDD) at least 2 units/day
* Weight ≥ 20 lbs
* HbA1c ≤ 10.5%
* For participants <18 years old, living with one or more parent/legal guardian knowledgeable about emergency procedures for severe hypoglycemia, present with the participant during and after the meal challenges, and willing to use the Dexcom Follow app (with push notifications turned on) for the duration of the study.
* For participants ≥18 years old, availability of a local contact who has access to the study participant, and willing to use the Dexcom Follow app (with push notifications turned on) for the duration of the study. If the participant lives alone, the local contact must live within 30 minutes and have access to the subject overnight.
* Investigator has confidence that the participant and/or parent/guardian can successfully operate all study devices and is capable of adhering to the protocol.
* Willing to use only aspart (novolog) or lispro (humalog) insulin with the study devices, with no use of long-acting basal insulin injections, or inhaled insulin with the study devices.
* Have current glucagon product to treat severe hypoglycemia (injectable or nasal) at home (site will provide prescription if they do not have one)
* Willing and able to perform study meal challenges.

Exclusion Criteria:

* More than 1 episode of diabetic ketoacidosis (DKA) in the past 6 months
* More than 1 episode of severe hypoglycemia (needing assistance) in the past 6 months
* Inpatient psychiatric treatment in the past 6 months
* For Female: Currently pregnant or planning to become pregnant during the time period of study participation

  1. A negative pregnancy test will be required for all females of child-bearing potential
  2. Counseling on appropriate birth control options will be provided to all females of child-bearing potential
* Concurrent use of any non-insulin glucose-lowering agent, other than metformin (for example, GLP-1 agonists, Symlin, DPP-4 inhibitors, SGLT-2 inhibitors, sulfonylureas).
* Hemophilia or any other bleeding disorder
* Hemoglobinopathy
* History of heart, liver, lung or kidney disease determined by investigator to interfere with the study
* History of allergic reaction to Humalog or Novolog
* Use of any medications determined by investigator to interfere with study
* Significant chronic kidney disease (which could impact CGM accuracy in investigator's judgment) or hemodialysis
* Concurrent use of any medication that could interfere with the study CGM, such as hydroxyurea
* History of adrenal insufficiency
* History of abnormal TSH consistent with hypothyroidism or hyperthyroidism that is not appropriately treated
* History of gastroparesis
* A condition, which in the opinion of the investigator or designee, would put the participant or study at risk
* Participation in another pharmaceutical or device trial at the time of enrollment or anticipated for during the time period of study participation
* Employed by, or having immediate family members employed by Tandem Diabetes Care, Inc., or having a direct supervisor at place of employment who is also directly involved in conducting the clinical trial (as a study investigator, coordinator, etc.); or having a first-degree relative who is directly involved in conducting the clinical trial

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Pinsker, MD, Study Director — Tandem Diabetes Care, Inc.
Locations (4):
- United States (4):
  - Barbara Davis Center (Pediatric Clinic), Aurora, Colorado
  - Barbara Davis Center, Aurora, Colorado
  - Joslin Diabetes Center, Boston, Massachusetts
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Brown SA, Laffel LM, Akturk HK, Forlenza GP, Shah VN, Wadwa RP, Cobry EC, Isganaitis E, Schoelwer M, Lu VS, Rueda R, Sherer N, Corbett JP, Sasson-Katchalski R, Pinsker JE. Randomized, Crossover Trial of Control-IQ Technology with a Lower Treatment Range and a Modified Meal Bolus Module in Adults, Adolescents, Children, and Preschoolers with Varying Levels of Baseline Glycemic Control. Diabetes Technol Ther. 2025 Mar;27(3):187-193. doi: 10.1089/dia.2024.0501. Epub 2024 Nov 26. PMID 39601043

RESULTS

PARTICIPANT FLOW:
Groups:
- Control-IQ 2.0 Lower Range First, Then Standard Range: After a 2 week Run-In Period with Control-IQ 1.5, participants will use t:slim X2 pump with Control-IQ technology 2.0 at a lower treatment range for two weeks, then at a standard treatment range for 2 weeks.
- Control-IQ 2.0 Standard Range First, Then Lower Range: After a 2 week Run-In Period with Control-IQ 1.5, participants will use t:slim X2 pump with Control-IQ technology 2.0 at a standard treatment range for two weeks, then at a lower treatment range for 2 weeks.
Period: Overall Study
Arm/Group | Control-IQ 2.0 Lower Range First, Then Standard Range | Control-IQ 2.0 Standard Range First, Then Lower Range
Started | 36 | 36
Completed | 36 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control-IQ 2.0 Lower Range First, Then Standard Range | Control-IQ 2.0 Standard Range First, Then Lower Range | Total
Number analyzed (Participants) | 36 | 36 | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.7 (14.2) | 16.3 (12.1) | 17.0 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 18 | 35
  Male | 19 | 18 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 3 | 10
  Not Hispanic or Latino | 29 | 32 | 61
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 32 | 32 | 64
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Severe Hypoglycemic Events
Description: Number of severe hypoglycemic events (with cognitive impairment such that assistance of another individual is needed for treatment) during study compared with data on severe hypoglycemic events reported by T1D Exchange clinic registry over a 3-month time period
Time Frame: 2 weeks
Measure: Number; unit: events
Groups:
- Lower Range; Standard Range: Participants will use t:slim X2 insulin pump with Control-IQ technology 2.0 with a lower range for two weeks.
Arm/Group | Lower Range | Standard Range
Number analyzed (Participants) | 72 | 72
events | 0 | 0

2. Primary Outcome: Number of Diabetic Ketoacidosis (DKA) Events
Description: Number of diabetic ketoacidosis during study compared with data on DKA events, compared with data on DKA events reported by T1D Exchange clinic registry over a 3-month time period
Time Frame: 2 weeks
Measure: Number; unit: events
Groups:
- Standard Range: Participants will use t:slim X2 insulin pump with Control-IQ technology 2.0 with a standard range for two weeks.
Arm/Group | Lower Range | Standard Range
Number analyzed (Participants) | 72 | 72
events | 0 | 0

3. Secondary Outcome: Percent of Time <54 mg/dL
Description: CGM percent time <54 mg/dL during each study period.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Lower Range | Standard Range
Number analyzed (Participants) | 72 | 72
percentage of time | 0.4 [0.1 to 0.8] | 0.3 [0.1 to 0.7]

4. Secondary Outcome: Percent of Time <70 mg/dL
Description: CGM percent time <70 mg/dL during each study period.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Lower Range | Standard Range
Number analyzed (Participants) | 72 | 72
percentage of time | 2.0 [0.9 to 3.3] | 1.6 [0.7 to 3.0]

5. Secondary Outcome: Percent Time 70-140 mg/dL
Description: CGM percent time 70-140 mg/dL during each study period.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Lower Range | Standard Range
Number analyzed (Participants) | 72 | 72
percentage of time | 43.9 [38.2 to 51.3] | 39.2 [30.9 to 48.1]

6. Secondary Outcome: Percent Time 70-180 mg/dL
Description: CGM percent time 70-180 mg/dL during each study period.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Groups:
- Control-IQ 2.0 Lower Range: Participants will use t:slim X2 pump with Control-IQ technology 2.0 at an Lower target for two weeks.
  t:slim X2 insulin pump with Control-IQ technology 2.0: t:slim X2 insulin pump with Control-IQ technology 2.0, and wearing the Dexcom G6 sensor.
Arm/Group | Lower Range | Control-IQ 2.0 Lower Range
Number analyzed (Participants) | 72 | 72
percentage of time | 68.0 [60.5 to 74.3] | 65.8 [54.4 to 73.0]

7. Secondary Outcome: Percent Time > 180 mg/dL
Description: CGM percent time >180 mg/dL during each study period.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Lower Range | Standard Range
Number analyzed (Participants) | 72 | 72
percentage of time | 30.5 [23.9 to 36.3] | 33.0 [25.2 to 43.8]

8. Secondary Outcome: Percent Time > 250 mg/dL
Description: CGM percent time >250 mg/dL during each study period.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Lower Range | Standard Range
Number analyzed (Participants) | 72 | 72
percentage of time | 9.9 [5.1 to 15.3] | 10.6 [5.7 to 18.5]

9. Secondary Outcome: Mean Glucose
Description: Mean CGM glucose mg/dL during each study period.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Lower Range | Standard Range
Number analyzed (Participants) | 72 | 72
mg/dL | 160.2 [149.7 to 172.6] | 166.0 [152.6 to 183.4]

10. Secondary Outcome: Glucose SD
Description: Glucose SD mg/dL during each study period.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Lower Range | Standard Range
Number analyzed (Participants) | 72 | 72
mg/dL | 63.5 [52.5 to 71.0] | 61.3 [53.8 to 72.7]

11. Secondary Outcome: Glucose Coefficient of Variation
Description: Glucose Coefficient of Variation (%) during each study period.
Time Frame: 2 weeks
Measure: Median (Inter-Quartile Range); unit: percentage of coefficient of variation
Arm/Group | Lower Range | Standard Range
Number analyzed (Participants) | 72 | 72
percentage of coefficient of variation | 38.1 [34.9 to 42.5] | 37.3 [34.0 to 41.4]

ADVERSE EVENTS:
Time Frame: Two weeks for each intervention.
Arm/Group | Lower Range | Standard Range
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/72
Other Adverse Events (participants affected / at risk) | 6/72 | 15/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lower Range (N=72) | Standard Range (N=72)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Hyperglycemia without ketosis (Endocrine disorders) | 2 (2) | 1 (1)
Hyperglycemia with ketosis (Endocrine disorders) | 1 (2) | 6 (6)
Foot Injury (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Yeast Infection (Infections and infestations) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1) — at site of CGM insertion
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 3 (3)
Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — at site of infusion set shortly after insertion
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Sprained Ankle (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-20): https://cdn.clinicaltrials.gov/large-docs/92/NCT05683392/Prot_SAP_000.pdf